CLINICAL TRIAL: NCT04536389
Title: Pregnancy Rates in Women With Normal Uterine Cavity With and Without Cervical Abnormalities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Momen Ahmed Mohammed Kamel, principle investigator, Assiut University
Other Study IDs: pearlstudy
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Intracytoplasmic Sperm Injection ,Hysteroscopicaly Detected Cervical Pathologies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: women with normal uterine cavity and normal cervix by office hysteroscopy.
  Interventions: Procedure: Office Hysteroscopy
- group B: women with normal uterine cavity with hysteroscopically detected cervical abnormality.
  Interventions: Procedure: Office Hysteroscopy

INTERVENTIONS:
Procedure: Office Hysteroscopy — The hysteroscope with its light source and flowing fluid was gently introduced into the vagina allowing for gradual distention. Once this was accomplished, the anatomy was followed with delicate movements. The hysteroscope was advanced under vision to the level of the ectocervix, and guided into the endocervical canal. Once the endocervical canal was completely explored, the endoscope was advanced across the internal cervical os to allow evaluation of the panoramic view of the uterine cavity.
  hysteroscopic correction of any detected lesion will be scheduled to the endoscopic operative list or the patient will receive the appropriate medical treatment.

SUMMARY:
The aim of our study is to investigate the pregnancy rates in women with normal uterine cavity ,with and without cervical abnormalities.

DETAILED DESCRIPTION:
The cervix is made up of the ectocervix and endocervix and is on average 3-4 cm long and 2.5 cm wide (Pardo et al., 2003; Mazouni et al., 2005; Robert et al., 2013). The ectocervix is the portion of the cervix projecting into the vagina. It is composed of non-keratinized stratified squamous epithelium and is divided into anterior and posterior lips. The squamocolumnar junction is the area where the epithelial cells of the endocervix and ectocervix meet (Herfs et al., 2013). In this area, the columnar cells of the endocervix undergo metaplasia to the squamous cells of the ectocervix. The opening of the ectocervix to the vagina is called the external os. Although studies of cervical length in non-pregnant women are few, it is acknowledged that the size and shape of both the cervix and the external os differ in women (Pardo et al., 2003; Mazouni et al., 2005) and vary with age, hormonal changes, parity and surgical treatments to the cervix.

Further evaluation of any cervical abnormalities by hysteroscopy eg. (choronic cervicitis , microcycstic epethelium ,micropolypi , cervical stenosis) before ICSI could address us to a hidden cause of infertility and may improve the pregnancy rates in ICSI cycles with prompt medical or surgical managment of such pathologies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women between 18 and 38 years old. 2. An indication for IVF/ICSI. 3. Women with primary or secondary infertility. 4. Women with BMI between 20 & 35.

Exclusion Criteria:

* 1. Refusal to join the study. 2. Untreated tubal hydrosalpinges. 3. Poor responders as assessed by AFC 4 or less, AMH O.8 ng/dl (nice 2013).

Ages: 18 Years to 38 Years | Sex: Female
Age Groups: Adult
Study Population: All infertile women will be assessed in IVF&ICSI unite of Women Health hospital,Assiut university and will be recruted according to the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 7thweek of prgnancy for cardiac pulsations
  clinical pregnancy rate will be described

SECONDARY OUTCOMES:
chemical pregnancy rate | 4 weeks
  chemical pregnancy rate will be described
Abortion rate | up to 28 weeks
  Abortion rate either first or second trimester abortion will be documented.
preterm labour | 9 months
  preterm labour will be described

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Women Health Hospital, Assiut University, Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pardo J, Yogev Y, Ben-Haroush A, Peled Y, Kaplan B, Hod M. Cervical length evaluation by transvaginal sonography in nongravid women with a history of preterm delivery. Ultrasound Obstet Gynecol. 2003 May;21(5):464-6. doi: 10.1002/uog.116. PMID 12768558
- [Result] Mazouni C, Bretelle F, Blanc K, Heckenroth H, Haddad O, Agostini A, Cravello L, Blanc B, Gamerre M. Transvaginal sonographic evaluation of cervix length after cervical conization. J Ultrasound Med. 2005 Nov;24(11):1483-6. doi: 10.7863/jum.2005.24.11.1483. PMID 16239649
- [Result] Robert AL, Nicolas F, Lavoue V, Henno S, Mesbah H, Poree P, Leveque J. [Ultrasonographic evaluation of the uterine cervix length remaining after LOOP-excision]. J Gynecol Obstet Biol Reprod (Paris). 2014 Apr;43(4):288-93. doi: 10.1016/j.jgyn.2013.03.014. Epub 2013 Apr 25. French. PMID 23623518
- [Result] Herfs M, Vargas SO, Yamamoto Y, Howitt BE, Nucci MR, Hornick JL, McKeon FD, Xian W, Crum CP. A novel blueprint for 'top down' differentiation defines the cervical squamocolumnar junction during development, reproductive life, and neoplasia. J Pathol. 2013 Feb;229(3):460-8. doi: 10.1002/path.4110. PMID 23007879